CLINICAL TRIAL: NCT01633424
Title: The "Stanford Integrated Psychosocial Assessment for Transplant" (SIPAT): Psychometric Characteristics of a New Scale for the Prediction of Post-transplant Psychosocial and Medical Outcomes.
Brief Title: The "Stanford Integrated Psychosocial Assessment for Transplant" (SIPAT)
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: CR-02
Record Dates: First submitted 2012-06-29; First posted 2012-07-04 (Estimated); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Organ Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Given the extremely limited availability of donated organs, transplant candidates must be carefully evaluated and selected to ensure the success of the transplant and value of the organ to the recipient. Medical criteria for pre-transplant evaluation of patients is well established, however, listing criteria for psychosocial risk factors (e.g., understanding of illness and transplant process, psychiatric history, support system, compliance, etc) is less standardized. The purpose of this research is to study the psychometric properties (e.g., predictive validity) of the new pre-transplant "Stanford Integrated Psychosocial Assessment for Transplant" (SIPAT) examination in patients who received heart, kidney, liver, or lung transplant and underwent the SIPAT evaluation before treatment. This new screening tool was designed to standardize the evaluation process of psychosocial risk factors and their severity, in order to enhance predictions of medical and psychosocial outcomes of patients post-transplant.

If the SIPAT is used for standard, pre-transplant assessment, risk factors that may be amenable to clinical intervention could be identified. In turn, this may assist in developing a comprehensive psychosocial treatment plan for each individual, with the ultimate goal of minimizing preventable problems, mitigating risk, and optimizing graft survival, patient function, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients identified through chart review who were transplanted with heart, kidney, liver, and lung between 6/1/2008 and 7/31/2011 and underwent the SIPAT evaluation before treatment.

Exclusion Criteria:

* Patients identified through chart review who were transplanted with heart, kidney, liver, and lung between 6/1/2008 and 7/31/2011, who did not undergo the SIPAT evaluation before treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 217 Stanford Hospital and Clinics patients fulfilled our criteria of being transplanted with heart, liver, kidney or lung between 6/1/2008 and 7/31/2011 and having been evaluated with SIPAT.
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Graft survival | Assessed at any given time post initial transplantation (up to 15 minutes to assess)
Patient survival | Assessed at any given time post initial transplantation (up to 15 minutes to assess)

CONTACTS AND LOCATIONS:
Overall Officials: José R. Maldonado, M.D., Principal Investigator — Stanford University
Locations (1):
- Stanford Hospitals and Clinics, Stanford, California, United States